CLINICAL TRIAL: NCT04729777
Title: Assessment of Cardiac Function Using Combined Cardiovascular Magnetic Resonance and Cardiopulmonary Exercise Testing (CMR-CPET)
Acronym: CMR-CPET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Actelion (Industry); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 100358; 226101 (Other: IRAS)
Record Dates: First submitted 2020-07-12; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Combined Cardiovascular Magnetic Resonance and Cardiopulmonary Exercise Testing — Clinical Cardiac MRI scan at rest with routine administration of gadolinium contrast agent. Participants then undergo the research component of the test which requires them to perform exercise, using a recumbent, MRI-compatible cycle ergometer, whilst their breathing is simultaneously analysed using a mask connected to a CPET machine, until they are limited by symptoms and they stop pedalling. Most participants will undergo only one scan. Some participants will be asked to have two or three such scans over 3 months to assess changes over time, and in response to standard treatment of pulmonary hypertension.

SUMMARY:
What problems limit patients' response to exercise? Using exercise cardiac magnetic resonance imaging to assess the heart's response, with simultaneous measurement of respiratory oxygen and carbon dioxide levels to assess the lung and skeletal muscle responses, to identify the rate-limiting factors affecting different types of patient

DETAILED DESCRIPTION:
Background and study aims Many medical conditions that affect the heart and lungs can cause breathlessness. People affected by breathlessness often require a number of tests to diagnose the medical condition responsible for their symptoms.

Cardiac MRI (magnetic resonance) scanning is already used to help diagnose and monitor patients with heart conditions (for example cardiomyopathy and pulmonary hypertension). By exercising while having an MRI scan, and at the same time measuring the gases breathed in and out from the air, it will be possible to more accurately understand the changes that occur in the heart, lungs and muscles.

The purpose of this study is to develop our understanding of the cardiovascular response to exercise in patients with non-ischaemic cardiomyopathy.

Who can participate? Patients aged 18 - 80 years with symptoms of breathlessness on exertion, and under the care of cardiology, pulmonary hypertension or rheumatology clinics for non-ischaemic cardiovascular disease.

What does the study involve? Participants will be invited to an appointment at the cardiovascular MRI department at the Royal Free Hospital. On the day of the appointment, participants will be welcomed to the department by the research team and the researchers will check that participants are well enough to exercise and safe to have an MRI scan. There will be an opportunity to ask any further questions.

The researchers will ask participants to perform exercise in one of three ways:

1. Using our special MRI safe exercise bike: The researchers will show participants how to use this and then the researchers will help participants to get on it and into the MRI scanner.
2. Lifting a weight using their arms: The researchers will check how much weight participants would be expected to manage before participants enter the scanner. The researchers will ask participants to lift and hold a weight using their dominant arm during the scan.
3. Stepping one (or both) leg(s) using an elastic resistance band. The researchers will measure the band so it is of the appropriate length for participants, and the researchers will show participants how to perform the exercise when in the scanner.

The researchers will give participants a special face mask to wear to measure the concentration of gases in exhaled breath (like carbon dioxide or oxygen) and breathing volumes. Most adults and children find the face mask comfortable and easy to wear.

The researchers will give participants a head-set so that participants can communicate at all times with the person running the scan.

First participants will have a MRI scan where the researchers ask participants to lie back and relax (this will take about 30 minutes).

Then the researchers will ask participants to exercise on the MRI safe bike for about 7 minutes, lift the weight for about 3 minutes, or perform leg stepping for about 3 minutes whilst participants are having continuous MRI scanning.

After the scan, the researchers will help participants out of the scanner.

What are the possible benefits and risks of participating? There are no individual benefits to taking part. The researchers hope that information from this study will help improve the understanding and treatment of heart conditions that can limit exercise ability. If participants like the researchers can make participants a copy of their scan on CD to keep. Sometimes the researchers might find new information that the researchers need to tell their treating doctor straight away. If the researchers do find such information the researchers will let participants and their doctor know as soon as possible. The researchers will reimburse reasonable travel expenses for participants to attend the research scan (unless participants are already scheduled to have a clinical visit on the same day). MRI scanning is very safe.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Symptoms of breathlessness on exertion under the care of cardiology, pulmonary hypertension or rheumatology clinics for non-ischaemic cardiovascular disease
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Previous ischaemic heart disease (including angina, myocardial infarction, PCI, CABG)
2. Unstable symptoms (including crescendo angina or angina at rest, and syncope on exercise)*
3. Arrhythmia**
4. Musculoskeletal disease preventing exercise
5. Patients unable to provide consent
6. General contraindications to CMR (e.g. implanted metal objects, pregnancy, severe claustrophobia)
7. Significant parenchymal lung disease (defined as >20% extent parenchymal disease on CT)
8. WHO functional class IV symptoms *Patients with unstable symptoms have been excluded as it would be unsafe for them to perform exercise whilst in a MRI scanner. Patients unable to exercise, WHO functional class IV and those with significant lung disease have been excluded as they would be unable to complete the exercise protocol **The researchers have excluded patients with arrhythmia as this can reduce the reliability of some of the CMR image sequences and also results in less predictable heart rate response to exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 - 80 years with symptoms of breathlessness on exertion, and under the care of cardiology, pulmonary hypertension or rheumatology clinics for non-ischaemic cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output (L/min) measured using aortic flow from PCMR measurements | Change from Baseline at 3 months
  Cardiac output (L/min) measured using aortic flow from PCMR measurements measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Ventricular volumes (mL) measured using volumetric measurements of both ventricles, at end-diastole and end-systole | Change from Baseline at 3 months
  Ventricular volumes (mL) measured using volumetric measurements of both ventricles, at end-diastole and end-systole measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Heart rate (bpm) from MRI ECG/heart rate monitor | Change from Baseline at 3 months
  Heart rate (bpm) from MRI ECG/heart rate monitor measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Blood pressure (mmHg) from MRI-compatible BP monitor | Change from Baseline at 3 months
  Blood pressure (mmHg) from MRI-compatible BP monitor measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Oxygen consumption (VO2, mL/min) from CPET machine | Change from Baseline at 3 months
  Oxygen consumption (VO2, mL/min) from CPET machine measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Carbon dioxide production (VCO2, mL/min) from CPET machine | Change from Baseline at 3 months
  Carbon dioxide production (VCO2, mL/min) from CPET machine measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Arteriovenous Oxygen Gradient (Muscle oxygen consumption, mlO2/100mL blood/min) calculated from Cardiac Output and VO2 | Change from Baseline at 3 months
  Arteriovenous Oxygen Gradient (Muscle oxygen consumption, mlO2/100mL blood/min) measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise calculated from Cardiac Output and VO2
Respiratory exchange ratio (RER) from CPET machine | Change from Baseline at 3 months
  Respiratory exchange ratio (RER) from CPET machine measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise
Exercise duration (sec) measured using a timer from the start to the end of exercise | Change from Baseline at 3 months
  Exercise duration (sec) measured using a timer from the start to the end of exercise measured at rest, at 2 minutes intervals during exercise, at 2 minutes and 4 minutes after end of exercise

SECONDARY OUTCOMES:
Cardiac Troponin T (ng/L) measured using blood sample prior to scan | through study completion, an average of 1 year
  Cardiac Troponin T (ng/L) measured using blood sample prior to scan and after scan
N-terminal pro-BNP (ng/L) measured using blood sample prior to scan | through study completion, an average of 1 year
  N-terminal pro-BNP (ng/L) measured using blood sample prior to scan and after scan
Haemoglobin (g/L) measured using blood sample prior to scan | through study completion, an average of 1 year
  Haemoglobin (g/L) measured using blood sample prior to scan and after scan
Autoantibody profile measured using blood sample prior to scan | through study completion, an average of 1 year
  Autoantibody profile measured using blood sample prior to scan and after scan
Invasive pulmonary pressures (PA systolic/diastolic/mean) in MR-RHC substudy measured using a pressure transducer at rest and after 1 min of exercise | through study completion, an average of 1 year
  Invasive pulmonary pressures (PA systolic/diastolic/mean) in MR-RHC substudy measured using a pressure transducer at rest and after 1 min of exercise
PH disease progression (WHO Functional class) measured using patient records | Change from baseline at 6 months
  PH disease progression (WHO Functional class) measured using patient records
Mortality measured using patient records | Change from baseline at 6 months
  Mortality measured using patient records

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data generated or analysed during this study will be included in the subsequent results publication